CLINICAL TRIAL: NCT00746135
Title: TRI-V Resynchronization in Paced Heart Failure Patients With ICD Indication.
Brief Title: TRI-V Heart Failure (HF) Implanted Cardioverter Defibrillator (ICD) Study
Acronym: TRI-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H37
Record Dates: First submitted 2008-08-20; First posted 2008-09-03 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
Keywords: Heart failure (NYHA class III and IV); Ventricular Dyssynchrony
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Conventional Biventricular Stimulation: RV Apex and LV Lead Tip
  Interventions: Device: Device Implantation
- B (Active Comparator): Anodal-Cathodal Biventricular Stimulation: cathodal LV Stimulation und anodal RVHis Stimulation = "Anodal-cathodal Bi-V".
  Interventions: Device: Device Implantation
- C (Active Comparator): Anodal-Cathodal Tri-V Stimulation: RV-apex and LV and RV-His
  Interventions: Device: Device Implantation

INTERVENTIONS:
Device: Device Implantation — RV apical pacing lead, RV pacing lead at HIS bundle position, LV pacing lead implantation
  Other Names: CRT-D Devices:; Atlas™ II+ HF / V-367 /St. Jude Medical; Epic™ II+ HF / V-357 / St. Jude Medical; Promote™ / 3207-36 / 3213-36 / St. Jude Medical; Adapters:; VIS 16 / Dr. Osypka GmbH

SUMMARY:
It's the aim of this study to investigate the impact of Right Ventricular (RV) lead position (RV-apex, His bundle area, RV-apex+His bundle area) in combination with individually optimized Left Ventricular (LV) lead placement and CRT timing on the outcome of cardiac resynchronization therapy (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Patient with indication for CRT-D: NYHA III-IV congestive heart failure, in spite of optimal medical treatment for their congestive heart failure
* LVEDD > 55 mm or > 30 mm/m² BSA
* EF < 35%
* Sinus rhythm and one of the following criteria:
* QRS >= 120 ms and PQ >= 200ms
* or
* 2nd / 3rd degree AV block
* Written informed consent

Exclusion Criteria:

* pacemaker indication (without ICD indication)
* tricuspidal valve and/or aortic valve replacement
* Indication for revascularization.
* less than 3 month after heart surgery or myocardial infarction
* hypertrophic obstructive cardiomyopathy
* intravenous catecholamine treatment
* uncorrected thyroid function
* severe kidney disorder (creatinin >2,5mg%)
* no written patient consent
* insufficient patient compliance
* participating in another study
* life expectancy < 1 year due to other severe disease
* age < 18 years
* no contraception (young women) or pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-11; Primary Completion 2010-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improvement according to Packer's "Heart Failure Clinical Composite Respond" | 12 months post implant

SECONDARY OUTCOMES:
Intraoperative Increase in Left Ventricular dp/dt | At Implant
Cardiopulmonary Capacity(Spiroergometry) | 12 months
Change in B-type natriuretic Peptide (BNP)-Concentration | 12 months
6 min walk test | 12 months
QoL assessment("Minnesota Living with Heart Failure = MLHF) | 12 months
12 channel ECG | 12 months
2D-echo optimized EF | 12 months
Complications and morbidity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kranig, MD, Principal Investigator — Departement of Cardiology - Electrophysiology- Heart Centre Osnabrück - Bad Rothenfelde
Locations (1):
- Departement of Cardiology - Electrophysiology- Heart Centre Osnabrück - Bad Rothenfelde, Bad Rothenfelde, Germany